CLINICAL TRIAL: NCT02553928
Title: Interventional, Randomised, Double-blind, Study to Evaluate the Safety and Tolerability of Once Daily Versus Twice Daily Memantine Treatment in Patients With Dementia of Alzheimer's Type and MMSE Range 5 - 18
Brief Title: Comparison of Once Daily and Twice Daily Dosing on Safety and Tolerability of Memantine in Patients With Alzheimer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14603A
Record Dates: First submitted 2015-09-16; First posted 2015-09-18 (Estimated); Results first posted 2019-03-14 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2018-11

CONDITIONS: Alzheimer Dementia (AD)
MeSH Terms: conditions — Alzheimer Disease | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Memantine (once daily) (Experimental): Memantine 20 mg once daily, tablets, orally AND Placebo tablets once daily, orally
  Interventions: Drug: Memantine (once daily)
- Memantine (twice daily) (Experimental): Memantine 10 mg twice daily, tablets, orally AND Placebo tablets twice daily, orally
  Interventions: Drug: Memantine (twice daily)

INTERVENTIONS:
Drug: Memantine (once daily)
  Other Names: Lu 00-800; Ebixa ®; Ebix ®
  Arms: Memantine (once daily)
Drug: Memantine (twice daily)
  Other Names: Lu 00-800; Ebixa ®; Ebix ®
  Arms: Memantine (twice daily)

SUMMARY:
Evaluation of the safety and tolerability of a 20 mg once daily dose of memantine compared with 10 mg given twice daily in patients with dementia of Alzheimer's type and MMSE range 5-18.

ELIGIBILITY:
Inclusion Criteria:

* The patient has a knowledgeable and reliable caregiver who will accompany the patient to all clinical visits during the study.
* The patient has a diagnosis of probable AD consistent with the National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria.
* The patient has a Mini Mental State Examination (MMSE) score ≥ 5 and ≤ 18 at Screening visit
* The dose of Memantine has been stable at 20 mg once a day for at least 3 month prior to screening

Exclusion Criteria:

* The patient has one or more of the following conditions: Evidence and/or history of any clinically significant neurodegenerative disease or other serious neurological disorders other than Alzheimer's disease including, but not limited to, Lewy body dementia, Fronto-Temporal dementia, Parkinson's disease, Huntington's disease, major cortical stroke, Multiple Sclerosis, major head trauma and primary or secondary cerebral neoplasm.
* The patient has a modified Hachinski ischemia score greater than 4 at the screening visit.
* The patient has any current psychiatric disorder or Axis I disorder (DSM-IV-TR™ criteria), established as the primary diagnosis, other than AD
* The patient is currently receiving treatment with an unstable dose of acetyl cholinesterase inhibitor

Other protocol defined inclusion and exclusion criteria may apply

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-10; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (6):
- China (6):
  - CN001, Beijing
  - CN006, Fujian
  - CN004, Shandong
  - CN002, Tianjin
  - CN007, Xi'an
  - CN003, Zhejiang

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Memantine (Once Daily) | Memantine (Twice Daily)
Started | 30 | 32
Completed | 28 | 29
Not Completed | 2 | 3
Not completed — Adverse Event | 2 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Administrative reason(s) | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Memantine (Twice Daily): 10 mg given twice daily, tablets, orally AND Placebo tablets twice daily, orally
- Total: Total of all reporting groups
Arm/Group | Memantine (Once Daily) | Memantine (Twice Daily) | Total
Number analyzed (Participants) | 30 | 32 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.1 (9.3) | 70.3 (8.1) | 69.7 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 34
  Male | 13 | 15 | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 30 | 32 | 62
MMSE Total Score [Mean (Standard Deviation); unit: units on a scale] — An 11-item test to assess cognitive aspects of mental function. Subtests assess orientation (item time, place), memory (item registration, recall), attention (item calculation), language (item naming assesses ability of naming, item repetition and comprehension assess the following of verbal commands, item reading assesses understanding of written commands, item writing assessed by writing a sentence spontaneously), and visual construction (item drawing). Scores are dichotomous for each item (1=correct response, 0=incorrect response). Total score=0-30; higher scores indicate lower deficit.
  units on a scale | 11.4 (4.2) | 11.4 (4.5) | 11.4 (4.3)
Modified Hachinski Ischemia Total Score [Mean (Standard Deviation); unit: units on a scale] — Hachinski Ischaemic Score is a tool helpful in the bedside differentiation of the commonest dementia types, dementia of Alzheimer's type (DAT) and vascular dementia (VaD). A cut-off score ≤4 for DAT and ≥7 for VaD has a sensitivity of 89% and a specificity of 89%(Moroney 1997). Modified Hachinski Ischemic Scale helps to differentiate between Alzheimer's type and multi-infarct dementia.Score can be 0 - 12. Lower score is more typical of a patient with Alzheimer's disease. Higher score is more typical for multi-infarct dementia.
  units on a scale | 1.6 (1.2) | 1.8 (0.9) | 1.7 (1.0)
Duration of Alzheimer's Disease [Mean (Standard Deviation); unit: years] | 2.1 (1.9) | 2.3 (1.9) | 2.2 (1.9)

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Number of patients who reported adverse events
Time Frame: baseline to week 16 (end of study)
Population: All patients treated
Measure: Count of Participants; unit: Participants
Arm/Group | Memantine (Once Daily) | Memantine (Twice Daily)
Number analyzed (Participants) | 30 | 32
Participants | 15 | 16

2. Secondary Outcome: ADCS - CGIC Score at Week 12
Description: The Alzheimer's Disease Cooperative Study - Clinical Global Impression of Change (ADCS-CGIC) is a semi-structured interview designed to assess clinically relevant changes in patients with Alzheimer's disease. Items in the ADCS-CGIC interview provide general information, and information about cognition, behaviour, social and daily functioning. Responses to ADCS-CGIC interview result in a global clinical judgement of severity (at baseline) and clinically relevant change at subsequent visits. Severity rated at baseline is only used for reference. The severity at baseline is rated on a 7-point Likert-type scale from 1(normal, not ill at all) to 7 (among the most extremely ill patients). The ADCS-CGIC relevant change is rated on a 7-point Likert-type scale from 1 (marked improvement) to 7 (marked worsening).
Time Frame: ADCS - CGIC score at Week 12
Population: Full analysis set - all randomised patients who took at least one dose of investigational medicinal product, and who had a valid baseline assessment and at least one valid post-baseline assessment of the ADCS-CGIC.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Memantine (Once Daily) | Memantine (Twice Daily)
Number analyzed (Participants) | 29 | 29
units on a scale | 3.92 (0.14) | 3.60 (0.14)
Statistical Analysis 1: Comparison: Memantine (Once Daily) vs Memantine (Twice Daily); The ADCS-CGIC was analyzed based on an analysis of covariance (ANCOVA) of ADCS-CGIC score at Week 12, with treatment and site as fixed factors, and baseline score as a covariate using observed cases; Test type: Other; p = 0.097, ANCOVA — Based on full analysis set; Mean Difference (Final Values) = 0.32, 95% CI 2-sided [-0.06 to 0.69], Standard Error of Mean 0.19 — The comparison is to BID memantine

ADVERSE EVENTS:
Time Frame: Baseline to week 16 (end of study)
Arm/Group | Memantine (Once Daily) | Memantine (Twice Daily)
Serious Adverse Events (participants affected / at risk) | 0/30 | 1/32
Other Adverse Events (participants affected / at risk) | 6/30 | 2/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Memantine (Once Daily) (N=30) | Memantine (Twice Daily) (N=32)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Memantine (Once Daily) (N=30) | Memantine (Twice Daily) (N=32)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 0 (0)
White blood cell count decreased (Investigations) | 2 (2) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No